CLINICAL TRIAL: NCT06453239
Title: Assessment the Diagnostic Value of Pro-Neurotensin as a Serum Biomarker in Metabolic Dysfunction-associated Steatotic Liver Disease
Brief Title: Assessment the Diagnostic Value of Pro-Neurotensin as a Serum Biomarker in MASLD
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Omnia Aboelwafa, MD, Sohag University
Other Study IDs: Soh-Med-24-04-05MD
Record Dates: First submitted 2024-06-05; First posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Steatosis of Liver
MeSH Terms: conditions — Fatty Liver

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- 40 adults categorized as MASLD patients
  Interventions: Diagnostic Test: Pro-Neurotensin level as a Serum Biomarker
- 40 adults of non-MASLD (controls)
  Interventions: Diagnostic Test: Pro-Neurotensin level as a Serum Biomarker

INTERVENTIONS:
Diagnostic Test: Pro-Neurotensin level as a Serum Biomarker — Pro-Neurotensin mediates the development of fatty liver disease. Neurotensin (NT) is a 13-amino acid peptide secreted by the neuroendocrine cells of the small intestine in response to fat ingestion, which facilitates fatty acid absorption through the gut in relation to food lipid content.

SUMMARY:
To assess the diagnostic significance of serum pro-NT in MASLD and ability to differentiate between early and advanced steatosis.

ELIGIBILITY:
Inclusion Criteria:

* Asymptomatic adults were randomly recruited from relatives of patients in Tropical Medicine and Gastroenterology Outpatient Clinic or the Inpatient Section of the department. Participants were categorized as MASLD patients if their abdominal US examination showed the criteria of fatty liver as described later or Non-MASLD (Controls) if they did not show these criteria.

Exclusion Criteria:

* (i) Patients aged <18 years or >75 years. (ii) History of Alcohol consumption. (iii) A diagnosis of liver diseases other than MASLD, including viral hepatitis, drug-induced liver injury, clinically suspected cases of autoimmune liver disease, Wilson's diseases, primary biliary cholangitis.

The control group had no illness to cause any inflammation; no usage of alcohol, drug, or herbal substances; no history of previous liver diseases; and was negative for viral hepatitis serology tests and had completely normal liver US.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A total of 80 asymptomatic adults will be randomly recruited from relatives of patients in Tropical Medicine and Gastroenterology outpatient clinic or the inpatient section of the department. Participants will be categorized as MASLD patients if their radiological investigation (By abdominal ultrasound examination and Fibroscan) shows the criteria of fatty liver (including 40 adults) or non-MASLD (controls) if they don't show these criteria (including 40 adults).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2024-07 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Assessment the Diagnostic Value of Pro-Neurotensin as a Serum Biomarker in Metabolic Dysfunction-associated Steatotic Liver Disease | Baseline
  To assess the diagnostic significance of serum pro-Neurotensin in metabolic dysfunction-associated steatotic liver disease and ability to differentiate between early and advanced steatosis.

CONTACTS AND LOCATIONS:
Overall Officials: Reem Mahmoud, lecturer, Study Director — Sohag

REFERENCES:
- [Background] Mohamed AA, Abo-Elmatty DM, Ezzat O, Mesbah NM, Ali NS, Abd El Fatah AS, Alsayed E, Hamada M, Hassnine AA, Abd-Elsalam S, Abdelghani A, Hassan MB, Fattah SA. Pro-Neurotensin as a Potential Novel Diagnostic Biomarker for Detection of Nonalcoholic Fatty Liver Disease. Diabetes Metab Syndr Obes. 2022 Jun 22;15:1935-1943. doi: 10.2147/DMSO.S365147. eCollection 2022. PMID 35769889
- [Background] Villar B, Bertran L, Aguilar C, Binetti J, Martinez S, Sabench F, Real M, Riesco D, Paris M, Del Castillo D, Richart C, Auguet T. Circulating Levels of Pro-Neurotensin and Its Relationship with Nonalcoholic Steatohepatitis and Hepatic Lipid Metabolism. Metabolites. 2021 Jun 10;11(6):373. doi: 10.3390/metabo11060373. PMID 34200577